CLINICAL TRIAL: NCT06230692
Title: Understanding the Influence of Diaphragm Structure and Function on the Control of Breathing During Exercise in Children
Brief Title: Diaphragm Structure and Function in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Simon Ho, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00108839
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Muscle Training
Keywords: Diaphragm; Control of Breathing; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inspiratory Muscle Training (IMT) (Experimental): Participants will be asked to perform inspiratory muscle training (breathing exercise) 5 days per week for 6 weeks at home.
  Interventions: Device: POWERbreathe Plus IMT

INTERVENTIONS:
Device: POWERbreathe Plus IMT — Inspiratory muscle training will be performed using the POWERbreathe Plus IMT (POWERbreathe International Ltd., Warwickshire, UK), a commercially available inspiratory pressure threshold device. In this type of training, airflow is occluded until the generated inspiratory pressure reaches the predetermined threshold, which can be set at increments of 8 cm H2O.
  During the first week of training, the target intensity will be set at 50% of baseline maximal inspiratory pressure (MIP.) During the second week, the target intensity will be set at 60% of baseline MIP. Beginning at the third week and for the remainder of the training program, the target intensity will be set at 75% of the participant's baseline MIP. The target volume will be 5 sets of 6 breaths per day (total of 30 breaths per day), separated by 1-minute rest breaks between sets. The frequency of training will be 5 days per week, for a duration of 6 weeks.

SUMMARY:
The purpose of this research is to study the feasibility of a specific training program for the breathing muscles (inspiratory muscle training) and the effects on how breathing is regulated during exercise in typically developing children.

DETAILED DESCRIPTION:
During the first study visit, participants will undergo a series of pulmonary function and muscle performance tests followed by treadmill walking trials at different speeds with concurrent expired gas analysis via a face mask. The participants will then perform a training program for the breathing muscles at home for 6 weeks. The research team will follow up each week via telehealth visits to support training. After the 6-week training program, participants will return in-person for a follow-up visit and will undergo the same series of assessments as the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Age range 6-12 years of age

Exclusion Criteria:

* History of neuromuscular, cardiac, or pulmonary disease
* Known intellectual or developmental problems that would preclude the ability to assent
* Ruptured eardrum
* Recent injury or condition (less than 6 months ago) that precludes strength testing or walking
* Recent (less than 2 weeks ago) or current respiratory or other type of illness

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent completion | 6 weeks
  Percentage of enrolled participants who complete the 6-week inspiratory muscle training protocol
Adherence to treatment protocol | 6 weeks
  Number of sets and repetitions of training breaths completed during the 6-week inspiratory muscle training protocol

SECONDARY OUTCOMES:
Maximal inspiratory pressure (measured in cm H2O) | 6 weeks
  Maximal pressure generated during an inspiratory maneuver, representing inspiratory muscle strength
Diaphragm thickness (measured in mm) | 6 weeks
  Thickness of the diaphragm muscle measured by noninvasive ultrasound imaging
Exercise ventilation | 6 weeks
  Ratio of ventilation to carbon dioxide production (VE/VCO2) during steady-state walking, representing ventilatory drive during exercise

OTHER OUTCOMES:
6-minute walk test distance (measured in m) | 6 weeks
  Maximal distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ho, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No